CLINICAL TRIAL: NCT03954028
Title: The Study on the Healing of Soft Tissue Augmentation by the Acellular Dermal Matrix and Autogenous Subepithelial Connective Tissue Graft
Brief Title: The Healing of Soft Tissue Augmentation by Acellular Dermal Matrix and Autogenous Subepithelial Connective Tissue Graft
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn with IRB
Sponsor: University of Florida (Other)
Collaborators: Dentsply Implants Manufacturing GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB201900963
Record Dates: First submitted 2019-04-26; First posted 2019-05-17 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Gingival Recession, Generalized; Graft Reaction
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: Patients needing gingival soft tissue augmentation will receive two kinds of gingival tissue graft material in a split-mouth design. The autogenous connective tissue (CTG) graft material will be randomized to apply to one half, and commercial acellular dermal matrix (ADM) materials will be used in the opposite half.
Who Masked: Investigator
Masking Description: The biopsy sites will be coded alphanumerically. The investigator performing the gingival grafts will be different from the examiner performing the gingival biopsies. The examiner performing the gingival biopsies will be blinded to the grafting type source of the biopsy sites.The results from coded samples will be reported to the PI, who will summarize the data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CTG Group (Active Comparator): Patients needing gingival soft tissue augmentation will receive two kinds of gingival tissue graft material in a split-mouth design. In this group, the autogenous connective tissue graft (CTG) material will be randomized to transplant to one side of the arch.
  Interventions: Procedure: Gingival Punch Biopsy after healing of Gingival Soft Tissue Augmentation
- ADM Group (Active Comparator): The patients needing gingival soft tissue augmentation will receive two kinds of gingival tissue graft material in a split-mouth design. In this group, the commercial acellular dermal matrix (ADM) materials will be transplanted to the opposite side of the arch with CTG transplants.
  Interventions: Procedure: Gingival Punch Biopsy after healing of Gingival Soft Tissue Augmentation

INTERVENTIONS:
Procedure: Gingival Punch Biopsy after healing of Gingival Soft Tissue Augmentation — Patients needing gingival soft tissue augmentation will receive two kinds of gingival tissue graft material in a split-mouth design. The autogenous connective tissue (CTG) graft material will be randomized to apply to one half, and commercial acellular dermal matrix (ADM) materials will be used in the opposite half. After 3 months of healing, a gingival punch biopsy will be performed in both sides to collect the tissues for analysis.

SUMMARY:
The study team proposes to prospectively compare the healing outcomes of autogenous soft tissue connective tissue graft (CTG) and Acellular dermis matrix (ADM) in a split-mouth design study for patients requiring modification of gingival soft tissue biotype. The researchers aim to investigate the earlier phase of graft healing after the grafting surgery by biopsy histology and by examining the alteration of gene profile during the healing of gingival tissue healing by molecular cell biological techniques.

DETAILED DESCRIPTION:
The investigators will perform a prospective clinical randomized controlled trial, and recruit 12 patients who need gingival soft tissue augmentation. It is a split-mouth design: CTG will be used in one side of soft tissue augmentation, and ADM will be used on the other side. 3 months after graft healing, clinical measurements including soft tissue thickness, transparency visualization, tissue profile record with impression cast study model, and digital photography of tissue will be performed. The gingival punch biopsies ( 2mm diameters) will be performed in both sides of grafting areas under the local oral anesthesia injection. The collected tissue will be split into two halves, one for histological examination, and another half for gene analysis.

ELIGIBILITY:
Inclusion Criteria:

* general healthy
* periodontal healthy (no PD >3mm, no BOP, no mobility at the test site and control site)
* patients identified need gingival biotype modification (need for increased tissue thickness) during the periodontal exam or referred from orthodontics

Exclusion Criteria:

* current smoker or smoking history
* taking Antibiotics or medicines within the last 3 months
* past history of gingival soft tissue augmentation/modification surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
The histological analysis of the gingival biopsy tissue. | Month 3---after the gingival biopsy procedures
  Histological analysis with standard coloration will assess the epithelium and underneath connective tissue within the gingival biopsy tissue. Signs of inflammation (ulcerations, infiltration of neutrophil cells, vessel structure) will be noted.

SECONDARY OUTCOMES:
The immunohistological analysis of the gingival biopsy. | Month 3---after the gingival biopsy procedures
  Immunohistological analysis using specific antibodies will locate the epithelium (collagen IV), the smooth muscle (Smooth muscle actin), and re-innvervation (protein gene product 9.5, calcitonin-related gene product) according to the similar study by Perotto, et al. 2017.
RT-qPCR analysis of gingival biopsy. | Month 3---after the gingival biopsy procedures
  The RT-qPCR analysis will measure the level of expression (compared to the housekeeping gene GAPDH) of RNA specific to the epithelium (collagen IV), the smooth muscle (Smooth muscle actin), re-innvervation (protein gene product 9.5, calcitonin-related gene product) and inflammation (IL-1, IL-6, MMP-8, TNF-alpha).

OTHER OUTCOMES:
change in the gingival biotype analysis before and after grafting surgery | Baseline; Month 3 (before the gingival grafting surgery and before the gingival biopsy which is 3 months after gingival grafting surgery)
  The gingival thickness measurement by visualization with periodontal probing, the soft tissue profile analysis with dental casts and digital photographs will be performed before the gingival grafting surgery and before the gingival biopsy which is 3 months after gingival grafting surgery.
The healing time of the gingival biopsy sites | Up to 7 days after gingival biopsy
  The gingival wound healing after biopsy will be compared between the sites

CONTACTS AND LOCATIONS:
Overall Officials: Jia Chang, DDS, MS, PhD, Principal Investigator — University of Florida College of Dentistry, Department of Periodontology

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data sets are to be shared include all collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available once the summary data are published.
Access Criteria: The PI will review requests and criteria for reviewing requests.

REFERENCES:
- [Background] McGuire MK, Scheyer ET. Randomized, controlled clinical trial to evaluate a xenogeneic collagen matrix as an alternative to free gingival grafting for oral soft tissue augmentation. J Periodontol. 2014 Oct;85(10):1333-41. doi: 10.1902/jop.2014.130692. Epub 2014 Mar 5. PMID 24597764
- [Background] Cummings LC, Kaldahl WB, Allen EP. Histologic evaluation of autogenous connective tissue and acellular dermal matrix grafts in humans. J Periodontol. 2005 Feb;76(2):178-86. doi: 10.1902/jop.2005.76.2.178. PMID 15974840
- [Background] de Resende DRB, Greghi SLA, Siqueira AF, Benfatti CAM, Damante CA, Ragghianti Zangrando MS. Acellular dermal matrix allograft versus free gingival graft: a histological evaluation and split-mouth randomized clinical trial. Clin Oral Investig. 2019 Feb;23(2):539-550. doi: 10.1007/s00784-018-2470-6. Epub 2018 Apr 30. PMID 29713889
- [Background] Menceva Z, Dimitrovski O, Popovska M, Spasovski S, Spirov V, Petrushevska G. Free Gingival Graft versus Mucograft: Histological Evaluation. Open Access Maced J Med Sci. 2018 Mar 27;6(4):675-679. doi: 10.3889/oamjms.2018.127. eCollection 2018 Apr 15. PMID 29731940
- [Background] Wei PC, Laurell L, Lingen MW, Geivelis M. Acellular dermal matrix allografts to achieve increased attached gingiva. Part 2. A histological comparative study. J Periodontol. 2002 Mar;73(3):257-65. doi: 10.1902/jop.2002.73.3.257. PMID 11922254
- [Background] Perotto S, Romano F, Cricenti L, Gotti S, Aimetti M. Vascularization and Innervation of Connective Tissue Grafts in the Treatment of Gingival Recessions: A Histologic and Immunohistochemical Study. Int J Periodontics Restorative Dent. 2017 Jul/Aug;37(4):551-558. doi: 10.11607/prd.3020. PMID 28609502